CLINICAL TRIAL: NCT01940536
Title: The Effect of Tranexamic Acid on Transfusion Rates in Intertrochanteric Hip Fractures: A Prospective, Double-Blind, Randomized Controlled Trial
Brief Title: The Effect of Tranexamic Acid on Transfusion Rates in Intertrochanteric Hip Fractures
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Possible change in study protocol
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13083
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Hip Fracture; Blood Loss
Keywords: Hip Fracture; Blood Transfusion; Blood Loss; Tranexamic Acid
MeSH Terms: conditions — Hip Fractures; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Active Comparator): 1g tranexamic acid, intravenous, at time of sudy enrollment and again a surgical incision
  Interventions: Drug: Tranexamic Acid
- Placebo Injection (Placebo Comparator): Placebo injection (normal saline) a time of study enrollment and again at time of surgical incision
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — antifibrinolytic
  Other Names: Cyclokapron
  Arms: Tranexamic Acid
Drug: Placebo — Placebo
  Arms: Placebo Injection

SUMMARY:
The goal of this study is to determine if the use of tranexamic acid, a safe and effective antifibrinolytic, in patients with intertrochanteric hip fractures will result in a reduction in blood transfusion rates. Treatment will be administered pre-operatively as well as at the time of surgical incision. The primary outcome will be need for blood transfusion. Secondary outcomes will include calculated perioperative blood loss, length of stay, cost of inpatient care, and rate of adverse events, including DVT, PE, infection, MI, cerebrovascular event, need for re-hospitalization or re-operation and 30 day mortality.

DETAILED DESCRIPTION:
All patients meeting specified criteria will be recruited for enrollment into the study. Informed consent will be obtained from the patient or health care proxy upon diagnosis of intertrochanteric hip fracture by the on-call orthopedic resident or research coordinator. At that time, each patient will be randomized into one of two cohorts (Figure 1) by the hospital's Investigational Pharmacy using computer generated randomization and allocation concealment. The Investigational Pharmacy will also be responsible for the storage, preparation and distribution of both the tranexamic acid and the placebo injections. The two patient groups will include:

1. 1g of intra-venous tranexamic acid upon presentation to the emergency department and again at the time of surgical incision.
2. Placebo injections upon presentation to the emergency department and again at the time of surgical incision.

Both patients and the treating surgeons will be blinded with regard to placebo vs. treatment until completion of the study. All patients will be treated surgically with a long trochanteric femoral nail (TFN). Blood transfusion criteria will remain consistent with hospital standards (Hb<8 g/dL or symptomatic anemia) as determined by an independent, blinded medical team who will follow the patient throughout the hospital stay. Total number of blood transfusions received will be documented upon patient discharge.

All patients will be permitted to weight bear as tolerated post-operatively and deep vein thrombosis (DVT) prophylaxis will be standardized: subcutaneous heparin, 5000 units every 8 hours beginning upon admission until 12 hours prior to surgery and beginning 6 hours after surgery for a total of 6 weeks. Calf mechanical compression devices will also be utilized during the inpatient stay and will remain on at all times with the exception of physical therapy sessions. Diagnostic studies to assess for thromboembolic events (i.e. DVT, pulmonary embolism (PE), and stroke) will be ordered only if the patient develops clinical signs or symptoms that justify their use. Patients will be followed at regular intervals (6wk, 3mo, 6mo, 1 year) and at each time point the patient will be asked to report any adverse events (DVT, PT, Stroke, myocardial infarction, infection, hospitalization) that have occurred since their last visit. In cases where patients are unable to accurately report their medical history, care providers will be questioned and records will be obtained from care facilities if necessary. An attempt will be made to contact any patient who is lost to follow-up via telephone and U.S. Mail.

Safety of the study will be monitored by an independent Data Safety Monitoring Board at 6 month intervals and the study will be discontinued at their discretion based on the number of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Intertrochanteric Hip Fracture
* Age >18

Exclusion Criteria:

* Preoperative use of anticoagulant (Clopidogrel, Warfarin, Enoxaparin, Fondaparinux, Rivaroxaban
* Allergy to Tranexamic Acid
* History of intracranial hemorrhage or significant GI or retroperitoneal bleed requiring hospitalization
* History of thromboembolic event (Stroke, Deep Vein Thrombosis, Pulmonary Embolism)
* History of cirrhosis or evidence of hepatic (AST/ALT >60) or renal dysfunction (Cr >1.5 or GFR <30)
* Coronary stents or prior diagnosis of CAD
* Color blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Blood transfusion rate | Hospital stay (3-7 days)

SECONDARY OUTCOMES:
Calculated Blood Loss | Hospial Stay (3-7 days)
Infection rate | 30-day
  Surgical site infection, Pneumonia, etc
Reoperation Rate | 1 year
Hospital Length of Stay | 30-day
  Length o acue hospitalization for initial injury and surgery
Myocardial Infarction | 1 year
Cost of acute care | 30-day
  Cost of initial hospital say and surgical intervention until initial discharge
DVT o Cerebrovascular Event | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dean G Lorich, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States

REFERENCES:
- [Derived] Gausden EB, Garner MR, Warner SJ, Levack A, Nellestein AM, Tedore T, Flores E, Lorich DG. Tranexamic acid in hip fracture patients: a protocol for a randomised, placebo controlled trial on the efficacy of tranexamic acid in reducing blood loss in hip fracture patients. BMJ Open. 2016 Jun 21;6(6):e010676. doi: 10.1136/bmjopen-2015-010676. PMID 27329438